CLINICAL TRIAL: NCT06478992
Title: A Multicenter Randomized Controlled Trial of Hysteroscopic Suture Fixation of Mirena in the Treatment of Adenomyosis
Brief Title: Hysteroscopic Suture Fixation of Mirena in the Treatment of Adenomyosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-20220610-0097-02
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Adenomyosis; Hysteroscopy
Keywords: Suture fixation; Expulsion; Mirena; Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the thickness of the thickest uterine myometrium ≥30mm (Other)
  Interventions: Procedure: A:hysteroscopic suture fixation of Mirena; Procedure: A: simple Mirena placement under hysteroscopy
- the thickness of the thickest uterine myometrium <30mm (Other)
  Interventions: Procedure: B: hysteroscopic suture fixation of Mirena; Procedure: B：simple Mirena placement under hysteroscopy

INTERVENTIONS:
Procedure: A:hysteroscopic suture fixation of Mirena — A(the thickness of the thickest uterine myometrium ≥30mm ):The Mirena is fixed to the uterine wall under hysteroscopy, and the endometrial tissue was routinely aspirated and scraped during the operation and sent for pathological examination.
  Arms: the thickness of the thickest uterine myometrium ≥30mm
Procedure: A: simple Mirena placement under hysteroscopy — A(the thickness of the thickest uterine myometrium ≥30mm):Mirena is routinely placed in the uterine cavity under hysteroscopy, and endometrial tissue was routinely aspirated and scraped during the operation and sent for pathological examination.
  Arms: the thickness of the thickest uterine myometrium ≥30mm
Procedure: B: hysteroscopic suture fixation of Mirena — B(the thickness of the thickest uterine myometrium<30mm):The Mirena is fixed to the uterine wall under hysteroscopy, and the endometrial tissue was routinely aspirated and scraped during the operation and sent for pathological examination.
  Arms: the thickness of the thickest uterine myometrium <30mm
Procedure: B：simple Mirena placement under hysteroscopy — B(the thickness of the thickest uterine myometrium<30mm):Mirena is routinely placed in the uterine cavity under hysteroscopy, and endometrial tissue was routinely aspirated and scraped during the operation and sent for pathological examination.
  Arms: the thickness of the thickest uterine myometrium <30mm

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of hysteroscopic Mirena fixation in patients with adenomyosis with enlarged uterus, compared with simple Mirena placement under hysteroscopy. Whether the curative effect is not inferior to and reduces the incidence of Mirena expulsion.

DETAILED DESCRIPTION:
This study was a multicenter, randomized (1:1 allocation to each group), double-blind, parallel controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Pain due to adenomyosis (lower abdominal pain and low back pain) visual analogue scale (VAS) ≥40mm or menstrual volume score (PBAC) ≥100;

  * Adenomyosis was confirmed by ultrasound or magnetic resonance imaging (MRI);

    * The uterine volume measured by transvaginal gynecological three-dimensional ultrasound was more than 150cm3 and less than 280cm3 (the volume was about 280cm3 at 10 weeks of pregnancy); ④ A strong desire to preserve the uterus; ⑤ No fertility requirements within nearly one year;

      * Premenopausal women aged ≥18 years old; ⑦ Willing and able to abide by the study protocol, and have the ability to clearly judge the amount of menstruation and the degree of pain.

Exclusion Criteria:

* Presence of contraindications to Mirena (known or suspected pregnancy, current pelvic inflammatory disease or recurrent pelvic inflammatory disease, lower genital tract infection, postpartum endometritis, infectious abortion within the past 3 months, cervicitis, cervical dysplasia, uterine or cervical malignant lesions, progestin-dependent tumors, abnormal uterine bleeding of unknown cause, congenital or acquired uterine abnormalities, these include fibroids that deform the cervix, conditions that increase susceptibility to infections, acute liver diseases or tumours, allergy to active ingredients or excipient);

  * Malignant tumors (including reproductive system and other systems);

    * Acute stage of heart, liver and kidney failure or other patients who cannot tolerate operation;

      * The history of Mirena displacement or expulsion;

        * Ultrasound showed the presence of ovarian chocolate cyst; ⑥ The presence of deep endometrial nodules by gynecological examination;

          * The presence of intramural or subserous myoma ≥3cm or any size of uterine submucosal myoma (type 0, 1, 2); ⑧ Patients who are unwilling to participate in the study or who were considered by the investigators to be unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
expulsion rate of the Mirena | 1, 3, 6, and 12 months postoperatively

SECONDARY OUTCOMES:
menstrual volume | 1, 3, 6, and 12 months postoperatively
dysmenorrhea | 1, 3, 6, and 12 months postoperatively
uterine size under ultrasound | 1, 3, 6, and 12 months postoperatively